CLINICAL TRIAL: NCT02597777
Title: Pilot Randomized Double-Blind Controlled Trial of Topical Acetyl Hexapeptide-8 and the Cosmetic Appearance of Oily Skin
Brief Title: Topical Acetyl Hexapeptide-8 and the Cosmetic Appearance of Oily Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 691537
Record Dates: First submitted 2015-10-31; First posted 2015-11-05 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Oily Skin
MeSH Terms: interventions — acetyl-glutamyl-glutamyl-methionyl-glutaminyl-arginyl-argininamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Side of face receiving placebo vehicle (Placebo Comparator): One half of the face (left or right side) will be randomized to receive the placebo lotion. Subjects will be asked to apply a pea-sized amount of the lotion to half of the face at twice daily application for 4 weeks.
  Interventions: Other: Placebo vehicle
- Side of face receiving AH8 lotion (Experimental): One half of the face (left or right side) will be randomized to receive the 10% Acetyl Hexapeptide-8 containing (AH8) lotion. Subjects will be asked to apply a pea-size amount of the lotion to the half of the face twice daily application for 4 weeks.
  Interventions: Other: Acetyl Hexapeptide-8

INTERVENTIONS:
Other: Acetyl Hexapeptide-8 — Acetyl-Hexapeptide-8 peptide solution will be diluted to a final concentration of 10% using Cetaphil facial lotion base
  Other Names: Argireline
  Arms: Side of face receiving AH8 lotion
Other: Placebo vehicle — Water will be diluted to a final concentration of 10% using Cetaphil facial lotion base.
  Arms: Side of face receiving placebo vehicle

SUMMARY:
This is a randomized double-blinded study examining the effect of topical Acetyl Hexapeptide-8 AH8) for improving the cosmetic appearance and experience of oily skin.

DETAILED DESCRIPTION:
The purpose of this randomized double-blinded study is to investigate whether topical Acetyl Hexapeptide-8 can improve oily skin. Up to 15 adult subjects will be recruited. Each half of the face will randomized to receive either topical treatment with AH8 10% Lotion formulated in Cetaphil® Moisturizing Facial Lotion or the placebo vehicle treatment consisting of Cetaphil® Moisturizing Facial Lotion only, at twice daily application for 4 weeks.

The study consists of a total of 3 sessions: baseline visit, and at 2 weeks and 4 weeks for follow up assessment. Subjects will also be asked to complete an Oily Skin Self-Assessment Scale (OSSAS) and an Oily Skin Impact Scale (OSIS) survey at the first session. They will be filling out two OSSAS surveys (one for each side of the face) at the second and third sessions. The OSSAS survey includes subjective assessment of four components of oily skin: visual, blotting, tactile, and sensation. At each visit, the cosmetic appearance the facial skin will be scored clinically by a dermatologist using a validated 3-point scale for shine (1 = high, 2, moderate or 3 = low), and oiliness (1 = normal, 2 = easily visible or 3 = extensive) 16. High-resolution digital photographs of the facial skin with the use of photography and facial analysis instrumentation will be taken at baseline and at each visit to document facial appearance and for image analysis of shine level. Sebum of the left and right cheeks will be measured by a sebumeter to correlate to the oily appearance noted on the high resolution facial photographs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18

Exclusion Criteria:

* Recent intradermal botulinum neurotoxin injection within the last 6 months.
* Known hypersensitivity to AH8
* Ablative resurfacing procedures to the face within 6 months of the study initiation
* Report of pregnancy or breastfeeding
* Use of immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Physician graded shine score | 4 weeks

SECONDARY OUTCOMES:
Patient satisfaction rated by each patient using the Oily Skin Self-Assessment Scale (OSSAS) | 2 week
Patient satisfaction rated by each patient using the Oily Skin Self-Assessment Scale (OSSAS) | 4 week
Assessment for local irritation from the topical emulsions | 4 weeks
  Secondary safety endpoint
Physician graded oiliness score | 2 weeks
Physician graded oiliness score | 4 weeks
Sebum measurement | 2 weeks
Sebum measurement | 4 weeks
Patient satisfaction rated by each patient using the Oily Skin Impact Scale (OSIS) | 2 weeks
Patient satisfaction rated by each patient using the Oily Skin Impact Scale (OSIS) | 4 weeks
Physician graded shine score | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, MS, CAT, Principal Investigator — University of California, Davis, Dermatology
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States